CLINICAL TRIAL: NCT06276205
Title: To Compare the Effectiveness of Vitamin D & Levothyroxine Combination Therapy and Levothyroxine Alone on Serum Lipid Profile in Patients With Hypothyroidism
Brief Title: Vitamin D & Levothyroxine Combination Versus Levothyroxine on Lipid Profile in Hypothyroidism
Acronym: ViDaLLiT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Sidrah Lodhi, Assistant Professor of Endocrinology, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1037/RC/KEMU
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hypothyroidism Primary; Lipid Disorder; Dyslipidemias
Keywords: levothyroxine; Vitamin D; Lipids; Hypothyroidism; Dyslipidemia
MeSH Terms: conditions — Hypothyroidism; Lipid Metabolism Disorders; Dyslipidemias | interventions — Vitamin D; Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D + Levothyroxine (Experimental)
  Interventions: Drug: Vitamin D; Drug: Levothyroxin
- Levothyroxine Alone (Active Comparator)
  Interventions: Drug: Levothyroxin

INTERVENTIONS:
Drug: Vitamin D — if Vitamin D level suboptimal, 50,000 IU/week for 8 weeks followed by 2000 IU/d
  if optimal Vitamin D level, 2000 IU/d
  Arms: Vitamin D + Levothyroxine
Drug: Levothyroxin — commenced at a dose of 1.6mcg/kg/day and will be titrated 8 weekly according to response
  Other Names: Thyroxine

SUMMARY:
The goal of this clinical trial is to study the improvement of lipid levels in hypothyroid individuals after staring treatment.

The main question it aims to answer is:

• whether adding Vitamin D to standard therapy has any additional benefits

Participants will be given Vitamin D in replacement doses according to their pre-existing Vitamin D level in addition to levothyroxine.

Researchers will compare them with another group receiving only levothyroxine to see how much lipids improve in them

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders.
* Age more than 12 years
* Biochemically hypothyroid (overt & subclinical)
* Vitamin D level between 10-70ng/ml
* TC <250mg/dl, LDL 70-144mg/dl, TGs 150-499mg/dl

Exclusion Criteria:

* Known Atherosclerotic Cardiovascular Disease
* BMI>35kg/m2
* History of Alcoholism (>14 units/day)
* History of Beta blocker intake
* Patient taking lipid lowering drugs

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Decline in Total Cholesterol | 24 weeks
  >9% decline from baseline
Decline in LDL | 24 weeks
  14% decline in LDL-C from baseline >14% decline from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan